CLINICAL TRIAL: NCT07073781
Title: A Double-blind Placebo-controlled Exploratory Trial to Assess the Impact of Daily Lab4P Probiotic Supplementation on Cognitive Performance and Metabolic Regulation in Overweight Young Adults With Impaired Glucose Regulation
Brief Title: Probiotic Impact on Cognitive Performance, and Metabolic Outcomes in Overweight Young Adults With Impaired Glucose Regulation
Acronym: ProCog
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leeds Beckett University (Other)
Collaborators: Cultech Ltd, Port Talbot, UK (Unknown)
Responsible Party: Principal Investigator, Lewis Hepburn, Principal Investigator, Leeds Beckett University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LBU-Lab4P-ProCogTrial-2025; i-NutriLife Hub PoC_R3_012 (Other Grant/Funding Number: Biotechnology and Biological Sciences Research Council (BBSRC) i-NutriLife Hub)
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Impaired Glucose Regulation; Impaired Glucose Tolerance (Prediabetes); Prediabetes (Insulin Resistance, Impaired Glucose Tolerance); Overweight (BMI > 25); Cognitive Dysfunction; Neurovascular Coupling Mechanism and Cognitive Function
Keywords: Probiotic supplementation; Psychobiotic; Cognitive performance; Metabolic function; Impaired glucose tolerance; Gut-brain axis
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State; Insulin Resistance; Overweight; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups (Lab4P or placebo) and will receive their assigned intervention daily for 12 weeks. There will be no crossover between groups, and outcomes will be assessed at multiple time points across the intervention period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving the Lab4P probiotic capsules (Experimental): Experimental group will consume oral dose of 50 billion Colony forming Units (CFU) once daily till delivery.
  Interventions: Dietary Supplement: Lab4p Probiotic Consortium
- Group receiving the identical, non-active placebo (Placebo Comparator): Microcrystalline cellulose/d each, up till delivery
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lab4p Probiotic Consortium — The investigational product in this study is Lab4P, a patented multi-strain probiotic consortium formulated as a food supplement and supplied in capsule form. Each daily dose contains a total of 5 × 10¹⁰ CFU of live bacteria, comprising five strains: Lactobacillus acidophilus CUL60 and CUL21, Lactobacillus plantarum CUL66, Bifidobacterium bifidum CUL20, and Bifidobacterium animalis subsp. lactis CUL34. In addition to probiotics, each capsule also contains three micronutrients at 100-200% of the recommended daily intake: Vitamin D (10 µg; 200%), Vitamin C (80 mg; 100%), and Zinc (10 mg; 100%).
  Lab4P is a marketed, human-approved product manufactured by Cultech Ltd. (Port Talbot, UK) and is classified as a food supplement, available for purchase without prescription. Both the active product and placebo will be identically packaged to maintain blinding.
  Arms: Group receiving the Lab4P probiotic capsules
Other: Placebo — Placebo capsules are composed of microcrystalline cellulose, and are identical in appearance to the test product.
  Arms: Group receiving the identical, non-active placebo

SUMMARY:
This 12-week, double-blind, placebo-controlled trial will examine whether daily supplementation with the Lab4P probiotic can improve cognitive performance and metabolic health in overweight adults aged 18 to 35 with impaired glucose tolerance, a preclinical condition where blood glucose regulation is mildly disrupted. Seventy participants will be randomly assigned to receive either Lab4P or a placebo. The study will assess changes in memory, executive function, and processing speed, along with blood glucose control, cardiovascular function, cholesterol levels, body composition, and markers of inflammation. The study will also analyse changes in the gut microbiome and evaluate the safety and tolerability of the probiotic.

DETAILED DESCRIPTION:
Global rates of Overweight and obesity are rising at unprecedented levels, contributing to increased metabolic disturbances such as impaired glucose metabolism. Disruptions in glucose regulation are both characteristic of and contributory to the pathogenesis of metabolic disorders, including type 2 diabetes (T2D). Clinical perturbations in glucose homeostasis are strongly associated with cognitive impairments, and an increased risk of neurodegenerative diseases. Increasing evidence suggests that even slightly impaired glucose metabolism (IGM) may contribute to cognitive decline.

Emerging evidence shows that cognitive impairments, including memory, executive function, and visuomotor deficits, can be observed in young adults with impaired glucose metabolism, alongside early markers of structural and functional brain changes. Neuroimaging studies have revealed reduced white matter integrity and decreased cerebral glucose metabolism in prediabetic individuals aged 22-35, particularly in brain regions associated with attention, self-regulation, and working memory.

These neurocognitive effects appear to be driven by early neurovascular unit (NVU) dysfunction, involving elevated blood glucose, insulin resistance (IR), endothelial damage, and inflammation. Exaggerated glucose excursions promote oxidative stress and impair endothelial function at the blood brain barrier, disrupting cerebral blood flow (CBF), glucose transport and metabolic homeostasis. Functional uncoupling between CBF and regional cerebral glucose metabolism has been directly observed in young adults with IR.

Together, these findings suggest that NVU dysfunction may underlie early cognitive decline in young adults with IGM, and that this population represents a critical target for early, non-pharmacological intervention. Probiotic formulations, including the probiotic consortium Lab4P, have shown promise in improving metabolic markers and reducing inflammation, with preclinical data suggesting potential cognitive and neuroprotective benefits. However, its procognitive effects in humans remain unexplored.

This trial will evaluate whether Lab4P supplementation can enhance cognitive performance, and cardiometabolic regulation in overweight young adults with IGM. By targeting a modifiable risk state early in life, the study aims to determine whether probiotic supplementation can serve as a viable strategy to mitigate long term neurocognitive and metabolic decline.

ELIGIBILITY:
Inclusion Criteria

* Aged 18-35 years
* Body Mass Index (BMI) between 25.0 and 29.9 kg/m² (classified as overweight)
* In good general health (self-reported)
* Normal self-reported sleep patterns, with no history of diagnosed sleep disorders
* Willing and able to provide informed consent
* Able to comply with study procedures, including fasting and oral glucose tolerance testing

Exclusion Criteria:

* Diagnosed diabetes (any type).
* Diagnosed sleep disorders.
* Fasting glucose >6.9 mmol/L during screening.
* History of bariatric surgery (e.g., gastric bypass, sleeve gastrectomy).
* Major surgery, significant illness, trauma, infection, or myocardial infarction within the past 6 weeks.
* Current use of medications affecting glucose metabolism or probiotics
* Pregnancy or actively trying to conceive
* Night shift work within the past month

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Verbal Memory Performance | Baseline to Week 12 (end of treatment).
  Assessed using the Cambridge Neuropsychological Test Automated Battery (CANTAB) Verbal Recognition Memory task (VRM) a computerized word list recall task, which measures accuracy in recalling previously presented verbal stimuli to evaluate verbal memory function.

SECONDARY OUTCOMES:
Visual Episodic Memory | Baseline to Week 12 (end of treatment).
  Measured using the Paired Associates Learning (PAL) task (CANTAB), which assesses the ability to remember the locations of visual patterns and form new associations.
Number of Participants Reporting One or More Adverse Events (AEs) or Serious Adverse Events (SAEs) | Baseline to Week 12 (end of treatment).
  All adverse events (AEs) and serious adverse events (SAEs) will be monitored through participant self-reports and case report forms. Events will be categorized by severity and relatedness to the study product.
Visuospatial Working Memory | Baseline to Week 12 (end of treatment).
  Measured using the Spatial Working Memory (SWM) task (CANTAB), which assesses the ability to temporarily retain and manipulate spatial information and use effective search strategies during problem-solving.
Executive function (Response Inhibition and Impulse Control) | Baseline to Week 12 (end of treatment).
  Measured using the Stop Signal Task (SST) (CANTAB), which assesses the ability to inhibit a dominant or preplanned motor response when signaled.
Executive function (Cognitive Flexibility and Attentional Set-Shifting) | Baseline to Week 12 (end of treatment).
  Measured using the Intra-Extra Dimensional Set Shift (IED) task (CANTAB), which assesses the ability to shift attention between different stimulus dimensions and adapt to changing rules. This evaluates cognitive flexibility and executive function.
Processing speed, Psychomotor Response, and Attention | Baseline to Week 12 (end of treatment).
  Measured using the Five Choice Reaction Time (RTI) task (CANTAB), which assesses how quickly and accurately participants respond to visual stimuli.
Cerebrovascular Reactivity (CVR) | Baseline to Week 12 (end of treatment).
  CVR reflects the ability of cerebral blood vessels to dilate or constrict in response to changes in carbon dioxide, indicating the health of the brain's vascular system. Measured via transcranial Doppler ultrasound of the middle cerebral artery in response to hypercapnia/hypocapnia challenge.
Flow-Mediated Dilation (FMD) | Baseline to Week 12 (end of treatment).
  Measured using ultrasound imaging of the brachial artery before and after a period of blood flow restriction using a pressure cuff. The artery's ability to dilate in response to the return of blood flow (reactive hyperemia) reflects endothelial function, an early indicator of vascular health and cardiovascular risk.
Global Sleep Quality | Baseline to Week 12 (end of treatment).
  Measured using the Pittsburgh Sleep Quality Index (PSQI) global score, a validated 19-item self-report instrument assessing subjective sleep quality over the past month.
Sleep Latency | Baseline to Week 12 (end of treatment).
  Assessed as a PSQI subcomponent, defined as the self-reported time (in minutes) taken to fall asleep on most nights.
Sleep Duration | Baseline to Week 12 (end of treatment).
  Assessed as a PSQI subcomponent, reflecting the average number of hours of sleep per night.
Sleep Efficiency | Baseline to Week 12 (end of treatment).
  Calculated as a PSQI subcomponent, defined as the ratio of total sleep time to time spent in bed, expressed as a percentage.
Sleep Disturbances | Baseline to Week 12 (end of treatment).
  Derived from PSQI items capturing the frequency of nocturnal awakenings and other sleep interruptions.
Sleep Medication Use | Baseline to Week 12 (end of treatment).
  Based on PSQI responses indicating frequency of pharmacological sleep aid use over the past month.
Daytime dysfunction | Baseline to Week 12 (end of treatment).
  Evaluated using PSQI items assessing difficulties staying awake during the day and maintaining enthusiasm for activities.
Glycated Haemoglobin (HbA1C) | Baseline to Week 12 (end of treatment).
  HbA1c reflects average blood glucose levels over the previous 2 to 3 months and is used to assess long-term blood sugar control. Measured from capillary blood using the Afinion 2 Analyzer (Abbott).
Fasting Blood Glucose | Baseline to Week 12 (end of treatment).
  This measure reflects short-term blood sugar levels and is used to assess baseline glucose regulation. Measured from capillary blood using an over-the-counter, CE-marked glucometer.
Glucose Tolerance (AUC) | Baseline to Week 12 (end of treatment).
  Assessed via a 2-hour oral glucose tolerance test (OGTT), with capillary blood glucose measured at 0, 30, 60, and 120 minutes post-glucose ingestion. These values will be used to calculate the area under the curve (AUC), which reflects how effectively the body regulates blood glucose over time.
Systolic blood pressure | Baseline to Week 12 (end of treatment).
  Measured using an automated oscillometric device (Omron). This measure reflects the pressure in the arteries when the heart contracts and is a key indicator of cardiovascular health.
Diastolic blood pressure | Baseline to Week 12 (end of treatment).
  Measured using an automated oscillometric device (Omron). This measure reflects the pressure in the arteries when the heart is at rest between beats and is an important marker of vascular function and cardiovascular risk.
Total Cholesterol | Baseline to Week 12 (end of treatment).
  Measured from a fasting capillary blood sample using the Cholestech LDX Analyzer (Abbott). This test provides total blood cholesterol levels, which are used to assess cardiovascular risk.
Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline to Week 12 (end of treatment).
  Measured from a fasting capillary blood sample using the Cholestech LDX Analyzer (Abbott). LDL-C contributes to plaque buildup in the arteries and is a key cardiovascular risk marker.
High-Density Lipoprotein Cholesterol (HDL-C) | Baseline to Week 12 (end of treatment).
  Measured from a fasting capillary blood sample using the Cholestech LDX Analyzer (Abbott). HDL-C helps remove excess cholesterol from the bloodstream and is protective against heart disease.
Triglycerides | Baseline to Week 12 (end of treatment).
  Measured from a fasting capillary blood sample using the Cholestech LDX Analyzer (Abbott). Triglycerides are a type of fat found in the blood and are used to assess metabolic health and cardiovascular risk.
Body Mass Index (BMI) | Baseline to Week 12 (end of treatment).
  Calculated as weight in kilograms divided by height in meters squared (kg/m²). Weight is measured using a calibrated digital scale and height with a stadiometer. BMI is a gold standard measure used to classify underweight, normal weight, overweight, and obesity.
Waist-to-Hip Ratio | Baseline to Week 12 (end of treatment).
  Calculated by dividing waist circumference by hip circumference. This ratio reflects fat distribution and is a marker of cardiometabolic risk.
Total Lean Mass | Baseline to Week 12 (end of treatment).
  Measured in kilograms using dual-energy X-ray absorptiometry (DXA). This measure reflects the total weight of muscle and other non-fat, non-bone tissues in the body.
Total Fat Mass | Baseline to Week 12 (end of treatment).
  Measured in kilograms using dual-energy X-ray absorptiometry (DXA). This reflects the total amount of fat tissue in the body.
Percent Body Fat | Baseline to Week 12 (end of treatment).
  Calculated from DXA-derived fat mass as a percentage of total body mass. This measure is used to evaluate body composition and excess adiposity-related risk.
Interleukin-6 (IL-6) | Baseline to Week 12 (end of treatment).
  Quantified from venous plasma samples using enzyme-linked immunosorbent assay (ELISA) kits. IL-6 is a pro-inflammatory cytokine associated with immune response and chronic inflammation.
Tumor Necrosis Factor-Alpha (TNF-α) | Baseline to Week 12 (end of treatment).
  Measured from venous plasma samples using ELISA kits. TNF-α is a cytokine involved in systemic inflammation and plays a role in metabolic and vascular dysfunction.
Gut Microbiota Diversity | Baseline to Week 12 (end of treatment).
  Assessed by 16S rRNA gene sequencing of DNA extracted from stool samples. Diversity will be measured using alpha diversity indices (e.g., Shannon Index), reflecting the richness and evenness of microbial communities.
Gut Microbiota Community Dispersion | Baseline to Week 12 (end of treatment).
  Assessed using beta diversity metrics such as Bray-Curtis dissimilarity and principal coordinates analysis (PCoA). This reflects variability in microbial composition between participants and time points.
Relative Abundance of Microbial Taxa | Baseline to Week 12 (end of treatment).
  Determined from 16S rRNA gene sequencing data by calculating the proportion of individual bacterial taxa present in stool samples. This measure assesses how specific microbial populations change over time.
Adherence Rate | Baseline to Week 12 (end of treatment).
  Assessed by capsule counts at the Week 12 visit and participant self-reports. The number of capsules taken will be calculated as a percentage of the total expected capsules over the 12-week intervention period.
Physical Discomfort Symptoms | Baseline to Week 12 (end of treatment).
  Assessed using a structured, self-administered questionnaire. Participants will indicate whether they experienced specific physical symptoms during the past 14 days, and on how many days each symptom occurred. Symptom categories include gastrointestinal (e.g., constipation, diarrhoea, bloating), systemic (e.g., sore throat, headache, muscle ache, cold symptoms), and medication or menstrual-related events (e.g., use of antibiotics, vaginal treatments, menstruation).

CONTACTS AND LOCATIONS:
Overall Officials: Lewis F Hepburn, Msc, Principal Investigator — Leeds Beckett University; Lauren Owen, PhD, Study Chair — Leeds Beckett University; Steve Trangmar, PhD, Study Chair — Leeds Beckett University
Locations (1):
- Leeds Beckett University, Leeds, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD collected during the trial will be shared. This includes outcome-level data related to cognitive performance, sleep quality, glucose regulation, lipid profiles, vascular function, inflammatory biomarkers, body composition, and gut microbiota composition.
Supporting Information: Study Protocol, ICF
Time Frame: IPD and supporting information will be available after publication of the primary trial results. Data will remain accessible for a minimum of 5 years following the end of the study or until the end of the institutional data retention period, whichever is longer.
Access Criteria: Access to IPD and supporting information will be granted to qualified researchers who provide a sound scientific rationale and appropriate ethical approvals. Requests will be evaluated by the study team and data custodians at Leeds Beckett University. Sensitive data will only be shared under a data-sharing agreement and subject to participant consent and ethics approval. Access will be coordinated via the Leeds Beckett University Thesis and Research Data Repository.
URL: https://libguides.leedsbeckett.ac.uk/research-support/symplectic-and-repositories/thesis-and-research-data-repository

REFERENCES:
- [Background] Zilliox LA, Chadrasekaran K, Kwan JY, Russell JW. Diabetes and Cognitive Impairment. Curr Diab Rep. 2016 Sep;16(9):87. doi: 10.1007/s11892-016-0775-x. PMID 27491830
- [Background] Webberley TS, Bevan RJ, Kerry-Smith J, Dally J, Michael DR, Thomas S, Rees M, Morgan JE, Marchesi JR, Good MA, Plummer SF, Wang D, Hughes TR. Assessment of Lab4P Probiotic Effects on Cognition in 3xTg-AD Alzheimer's Disease Model Mice and the SH-SY5Y Neuronal Cell Line. Int J Mol Sci. 2023 Feb 28;24(5):4683. doi: 10.3390/ijms24054683. PMID 36902113
- [Background] Sadler JR, Shearrer GE, Burger KS. Alterations in ventral attention network connectivity in individuals with prediabetes. Nutr Neurosci. 2021 Feb;24(2):140-147. doi: 10.1080/1028415X.2019.1609646. Epub 2019 Apr 28. PMID 31030631
- [Background] Ribeiro M, Yordanova YN, Noblet V, Herbet G, Ricard D. White matter tracts and executive functions: a review of causal and correlation evidence. Brain. 2024 Feb 1;147(2):352-371. doi: 10.1093/brain/awad308. PMID 37703295
- [Background] Repple J, Karliczek G, Meinert S, Forster K, Grotegerd D, Goltermann J, Redlich R, Arolt V, Baune BT, Dannlowski U, Opel N. Variation of HbA1c affects cognition and white matter microstructure in healthy, young adults. Mol Psychiatry. 2021 Apr;26(4):1399-1408. doi: 10.1038/s41380-019-0504-3. Epub 2019 Aug 29. PMID 31467393
- [Background] Nazaribadie M, Amini M, Ahmadpanah M, Asgari K, Jamlipaghale S, Nazaribadie S. Executive functions and information processing in patients with type 2 diabetes in comparison to pre-diabetic patients. J Diabetes Metab Disord. 2014 Feb 4;13(1):27. doi: 10.1186/2251-6581-13-27. PMID 24495302
- [Background] Michael DR, Davies TS, Jack AA, Masetti G, Marchesi JR, Wang D, Mullish BH, Plummer SF. Daily supplementation with the Lab4P probiotic consortium induces significant weight loss in overweight adults. Sci Rep. 2021 Jan 6;11(1):5. doi: 10.1038/s41598-020-78285-3. PMID 33408364
- [Background] Lamport DJ, Lawton CL, Mansfield MW, Dye L. Impairments in glucose tolerance can have a negative impact on cognitive function: a systematic research review. Neurosci Biobehav Rev. 2009 Mar;33(3):394-413. doi: 10.1016/j.neubiorev.2008.10.008. Epub 2008 Nov 5. PMID 19026680
- [Background] Kullmann S, Heni M, Hallschmid M, Fritsche A, Preissl H, Haring HU. Brain Insulin Resistance at the Crossroads of Metabolic and Cognitive Disorders in Humans. Physiol Rev. 2016 Oct;96(4):1169-209. doi: 10.1152/physrev.00032.2015. Epub 2016 Aug 3. PMID 27489306
- [Background] Kirvalidze M, Hodkinson A, Storman D, Fairchild TJ, Bala MM, Beridze G, Zuriaga A, Brudasca NI, Brini S. The role of glucose in cognition, risk of dementia, and related biomarkers in individuals without type 2 diabetes mellitus or the metabolic syndrome: A systematic review of observational studies. Neurosci Biobehav Rev. 2022 Apr;135:104551. doi: 10.1016/j.neubiorev.2022.104551. Epub 2022 Jan 29. PMID 35104494
- [Background] Feng L, Gao L. The role of neurovascular coupling dysfunction in cognitive decline of diabetes patients. Front Neurosci. 2024 Mar 21;18:1375908. doi: 10.3389/fnins.2024.1375908. eCollection 2024. PMID 38576869
- [Background] Di Pino A, Urbano F, Scicali R, Di Mauro S, Filippello A, Scamporrino A, Piro S, Purrello F, Rabuazzo AM. 1 h Postload Glycemia Is Associated with Low Endogenous Secretory Receptor for Advanced Glycation End Product Levels and Early Markers of Cardiovascular Disease. Cells. 2019 Aug 16;8(8):910. doi: 10.3390/cells8080910. PMID 31426413
- [Background] Deery HA, Liang E, Di Paolo R, Voigt K, Murray G, Siddiqui MN, Egan GF, Moran C, Jamadar SD. The association of regional cerebral blood flow and glucose metabolism in normative ageing and insulin resistance. Sci Rep. 2024 Jun 25;14(1):14574. doi: 10.1038/s41598-024-65396-4. PMID 38914735
- [Background] Deery HA, Liang E, Di Paolo R, Voigt K, Murray G, Siddiqui MN, Egan GF, Moran C, Jamadar SD. Peripheral insulin resistance attenuates cerebral glucose metabolism and impairs working memory in healthy adults. NPJ Metab Health Dis. 2024 Aug 2;2(1):17. doi: 10.1038/s44324-024-00019-0. PMID 40604159

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT07073781/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT07073781/ICF_001.pdf